CLINICAL TRIAL: NCT00162942
Title: A Randomized, Prospective, Double-Blinded, Placebo-Controlled (Sham-Controlled) Study to Evaluate the Safety and Effectiveness of the Adacolumn Apheresis System for the Treatment of Moderate to Severe Crohn's Disease
Brief Title: Study for the Treatment of Crohn's Disease With Adacolumn
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka America Pharmaceutical (Industry)
Responsible Party: Tao Wang / Director of Medical Affairs, Otsuka America Pharmaceutical, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 512-04-206
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Results first posted 2009-04-07 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Adacolumn (Active Comparator): Adacolumn, ten apheresis sessions within 9 weeks
  Interventions: Device: Adacolumn
- Sham (Sham Comparator): Sham, ten apheresis sessions within 9 weeks
  Interventions: Device: Sham

INTERVENTIONS:
Device: Adacolumn — Ten apheresis sessions:
  One hour of Adacolumn Apheresis System procedure per visit. Patient had two procedures per week for the first two weeks followed by one apheresis session per weeks for two weeks (Weeks 1-4). then a week break occurs for rest followed by one apheresis session per week for 4 weeks (weeks 6-9).
  Arms: Adacolumn
Device: Sham — Sham, ten apheresis sessions within 9 weeks
  Arms: Sham

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Adacolumn Apheresis System as a treatment for the signs and symptoms of Crohn's disease.

DETAILED DESCRIPTION:
Trial Features:

* Medical device (Non-drug option)
* Most patients can remain on current treatment regimen throughout the study

Components of the Study:

* Study length is 24 weeks, which includes a screening visit, ten treatment visits over nine weeks and 4 follow-up appointments
* Physical exams, laboratory tests and disease assessments conducted at no charge to the patient
* 2:1 Randomization (treatment:sham)
* Open-Label extension offered to eligible patients

ELIGIBILITY:
Key Inclusion Criteria:

* Moderate to severe Crohn's disease
* Adequate peripheral venous access
* Agree to participate in the required follow-up visits
* Able to complete a diary
* Signed written informed consent document and authorization for use of protected health information

Key Exclusion Criteria:

* Extremely severe Crohn's disease
* Known obstructive symptoms within the past 3 months
* Presence of toxic megacolon
* Major surgery within the past 6 weeks or anticipated need for surgery within 12 weeks
* Total colectomy, ileostomy, stoma or 100 cm of resected small bowel
* Requiring in-patient hospitalization
* A history of allergic reaction to heparin or heparin-induced thrombocytopenia
* A history of hypersensitivity reaction associated with an apheresis procedure or intolerance of apheresis procedures
* A history of severe cardiovascular or peripheral arterial diseases
* A history of cerebral vascular diseases
* Liver diseases
* Renal insufficiency
* Known bleeding disorder or use of concomitant anticoagulant therapy for purposes other than apheresis treatment
* Any hypercoagulable disorder
* Known infection with Hepatitis B or C, or HIV
* Severe anemia
* Leukopenia or granulocytopenia
* Evidence of current systemic infection
* Malignancy
* Pregnant, lactating or planning to become pregnant during the course of the investigational study
* Used within the last 30 days, an investigational drug, biologic or device or 5 half-lives, if known, for any investigational drug or biologic

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yosuke Komatsu, MD, PhD, Study Director — Otsuka America Pharmaceutical
Locations (36):
- United States (28):
  - Mayo Clinic Scottsdale, Phoenix, Arizona
  - Capitol Gastroenterology Consultants Medical Group, Roseville, California
  - UCSF Mount Zion Medical Center, San Francisco, California
  - Rocky Mountain Gastroenterology Associates, PC, Wheat Ridge, Colorado
  - Medical Research Institute of Connecticut, Hamden, Connecticut
  - Venture Research Institute, LLC, North Miami Beach, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Metropolitan Gastroenterology Group, Chevy Chase, Maryland
  - Massachusetts General Hospital, GI Unit, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, Clinton Township, Michigan
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Long Island Clinical Research Associates, Great Neck, New York
  - University of North Carolina, Division of Digestive Disease & Nutrition, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Columbia Gastroenterology Associates, Columbia, South Carolina
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Washington Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Madison, Wisconsin
  - University of Wisconsin-Madison, Madison, Wisconsin
- Canada (8):
  - Walter Mackenzie Health Sciences Centre, Edmonton, Alberta
  - Gastroenterology & Hematology Clinic, Abbotsford, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Hotel-Dieu Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Sands BE, Katz S, Wolf DC, Feagan BG, Wang T, Gustofson LM, Wong C, Vandervoort MK, Hanauer S. A randomised, double-blind, sham-controlled study of granulocyte/monocyte apheresis for moderate to severe Crohn's disease. Gut. 2013 Sep;62(9):1288-94. doi: 10.1136/gutjnl-2011-300995. Epub 2012 Jul 3. PMID 22760005

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adacolumn | Sham
Started | 157 | 78
Week 12 | 127 | 61
Completed | 51 | 26
Not Completed | 106 | 52
Not completed — Adverse Event | 10 | 6
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Physician Decision | 1 | 0
Not completed — Enter Open-Label Study | 76 | 35
Not completed — Alternate Therapy | 6 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Flare During Active Treatment | 7 | 3
Not completed — 2 or more consecutive treatments missed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adacolumn | Sham | Total
Number analyzed (Participants) | 157 | 78 | 235
Age Continuous [Mean (Standard Deviation); unit: years] | 40.6 (12.5) | 41.4 (13.6) | 40.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 44 | 125
  Male | 76 | 34 | 110
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 142 | 75 | 217
  Hispanic | 2 | 0 | 2
  African American | 8 | 2 | 10
  Asian/Pacific Islander | 1 | 0 | 1
  Other | 4 | 1 | 5
Alcohol Use [Number; unit: participants]
  Consumes Alcohol | 85 | 54 | 139
  Previously Drank | 33 | 12 | 45
  Never Drank | 39 | 12 | 51
Smoking Status [Number; unit: participants]
  Current Smoker | 46 | 26 | 72
  Ex-Smoker | 39 | 23 | 62
  Non-Smoker | 72 | 29 | 101
Baseline Crohn's Disease Activity Index Score [Mean (Standard Deviation); unit: units on a scale] — 601-point, ordinal scale which quantifies the symptoms of patients with Crohn's Disease from 0 (complete remission) to 600 (most severe active disease)
  units on a scale | 309.6 (55.7) | 314.7 (53.5) | 311.3 (54.9)
Crohn's Disease History [Mean (Standard Deviation); unit: months] — Time, since diagnosis of Crohn's Disease, was collected at baseline.
  months | 139.5 (125.1) | 129.9 (123.1) | 136.3 (124.3)
Height [Mean (Standard Deviation); unit: centimeter] | 170.3 (9.7) | 169.9 (10.3) | 170.2 (9.9)
Inflammatory Bowel Disease Flares in the Past 12 Months [Mean (Standard Deviation); unit: flares] | 2.2 (2.2) | 2.5 (2.8) | 2.3 (2.4)
Weight [Mean (Standard Deviation); unit: kilogram] | 74.89 (16.22) | 72.29 (19.23) | 74.03 (17.28)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Remission
Description: Clinical Remission is defined as a Crohn's Disease Activity Index (CDAI) score of ≤150 when evaluated at Week 12
Time Frame: Baseline to Week 12
Population: All subjects who received at least one apheresis treatment session were included in the intent-to-treat population (ITT). The ITT was used for effectiveness analysis. The week 12 CDAI score was used for the analysis. Subjects without a week 12 CDAI score or with a major violation on prohibited medications were considered a treatment failure.
Measure: Number; unit: percentage of participants
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 157 | 78
percentage of participants | 17.8 | 19.2
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = .858, Fisher Exact

2. Primary Outcome: Frequency and Severity of Adverse Events Through Week 12
Description: All subjects who received at least one apheresis treatment session were included in the intent-to-treat population (ITT). The ITT population was used for effectiveness analysis.
Time Frame: Baseline through Week 12 Visit
Population: All subjects who received at least one apheresis treatment session were included in the intent-to-treat population (ITT). The ITT population was used for effectiveness analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 157 | 78
percentage of participants
  Any Adverse Event | 93 | 93.6
  Severe Adverse Event | 19.7 | 19.2
  Device-Related Adverse Event | 61.1 | 75.6
  Serious Adverse Event | 8.3 | 6.4
  Device-Related Serious Adverse Event | 0.6 | 0.0
  Adverse Event Leading to Device Discontinuation | 10.8 | 11.5

3. Secondary Outcome: CDAI Score Change From Baseline
Description: 601-point, ordinal scale which quantifies the symptoms of patients with Crohn's Disease from 0 (complete remission) to 600 (most severe active disease). Mean change=Week 12 Mean CDAI-Baseline Mean CDAI
Time Frame: Baseline to Week 12
Population: All subjects who received at least one apheresis treatment session were included in the intent-to-treat population (ITT). The ITT population was used for effectiveness analysis. The week 12 score was used for the analysis. If no week 12 score, then the week 9 score was be used. If no week 9 score, the subject was considered a treatment failure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 152 | 73
units on a scale | -65.6 (96.6) | -62.3 (103)
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.813, Student's t-test

4. Secondary Outcome: Clinical Response
Description: Clinical Response is defined as a ≥ 100-point reduction in the CDAI scores at Week 12
Time Frame: Baseline to Week 12
Population: All subjects who received at least one apheresis session were included in the intent-to-treat population (ITT). The ITT population was used for effectiveness analysis. The week 12 CDAI score or Last Observation Carried Forward was used for the analysis. Subjects with a major violation on prohibited medications were considered a treatment failure.
Measure: Number; unit: percentage of participants
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 157 | 78
percentage of participants | 28.0 | 26.9
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 1.000, Fisher Exact

5. Secondary Outcome: Mean Change in Short-Form 36 Questionnaire (SF-36) Physical Component Summary (PCS) Score
Description: 101-point, ordinal scale measuring general health of patients from 0 (low quality of life) to 100 (high quality of life), Mean change=Week 12 Mean -Baseline Mean
Time Frame: Baseline to Week 12
Population: All subjects who received at least one apheresis treatment session were included in the intent-to-treat population (ITT). The ITT population was used for effectiveness analysis. The week 12 score or Last Observation Carried Forward was used for the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 145 | 71
units on a scale | 3.84 (8.76) | 3.29 (9.19)
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.670, Student's t-test

6. Secondary Outcome: Mean Change in Short-Form 36 Questionnaire (SF-36) Mental Component Summary (MCS) Score
Description: as for outcome 5
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 145 | 71
units on a scale | 2.52 (10.13) | 2.48 (11.23)
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.977, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Mean Change in Inflammatory Bowel Diseases Questionnaire (IBDQ)
Description: 193-point, ordinal scale measuring disease-specific quality of life from 32 (low quality of life) to 224 (high quality of life). Mean change= Week 12 Mean-Baseline Mean
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 148 | 74
units on a scale | 18.5 (32.1) | 16.8 (37.9)
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.670, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Mean Change in EuroQol Score (Single Index)
Description: A continuous scale that is a cardinal index of health from 0 (no impairment) to 1 (most impairment), Mean change=Week 12 Mean -Baseline Mean
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 147 | 72
units on a scale | 0.0392 (0.2239) | 0.0917 (0.2648)
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.170, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Mean Change in EuroQol Score (Visual Analog Scale)
Description: 101-point, ordinal scale which measures non-disease specific health-related quality of life from 0 (Worst imaginable health state) to 100 (best imaginable health state)
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 148 | 73
units on a scale | 4.4 (19.8) | 5.5 (18.6)
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.0773, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Mean Change in Work Limitations Questionnaire (Time Management)
Description: 101-point, ordinal scale which measures the degree to which health problems interfere with certain aspects of job performance and productivity from 0 (limited none of the time) to 100 (limited all the time), Mean change=Week 12 Mean -Baseline Mean
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 132 | 63
units on a scale | -9.9 (25.5) | -6.6 (31.7)
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.261, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Mean Change in Work Limitations Questionnaire (Physical Demands)
Description: as for outcome 10
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 136 | 68
units on a scale | -5.2 (23.1) | 2.3 (22.7)
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.379, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Mean Change in Work Limitations Questionnaire (Mental-Interpersonal Demands)
Description: as for outcome 10
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 136 | 66
units on a scale | -5.5 (20.5) | -2.7 (20.8)
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.441, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Mean Change in Work Limitations Questionnaire (Output Demands)
Description: as for outcome 10
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 132 | 63
units on a scale | -7.4 (25.8) | -3.8 (28.7)
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.759, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Mean Change in Work Limitations Questionnaire (WLQ Index)
Description: as for outcome 10
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 123 | 59
units on a scale | -1.8 (5.6) | -0.5 (6.9)
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.222, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Mean Change in Crohn's Disease Endoscopic Index of Severity
Description: 26-point,ordinal scale that assesses the severity of Crohn's Disease from 0 (least severe) to 26 (most severe), Mean change=Week 12 Mean -Baseline Mean
Time Frame: Baseline to Week 12
Population: Endoscopic evaluations were to be performed at baseline and Week 12 on a subset of study subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 25 | 8
units on a scale | 2 (7.73) | -4.63 (13.20)
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.256, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Mean Change in Subject Global Rating
Description: 7-point,ordinal scale that measures the subject's state of Crohn's Disease from 0 (totally inactive) to 7 (as bad as it gets), Mean change=Week 12 Mean -Baseline Mean
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 149 | 71
units on a scale | -0.7 (1.6) | -0.6 (1.3)
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.870, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Mean Change in C-Reactive Protein
Time Frame: Baseline to week 12
Population: All subjects who received at least one apheresis treatment session were included in the intent-to-treat population (ITT). The ITT population was used for effectiveness analysis. The week 12 value or Last Observation Carried Forward was used for the analysis.
Measure: Mean (Standard Deviation); unit: milligrams/liter
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 147 | 71
milligrams/liter | -1.75 (22.67) | 0.24 (12.59)
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.350, Wilcoxon (Mann-Whitney)

18. Post Hoc Outcome: Clinical Response in Subjects With a CDAI Score Greater Than 300
Description: A clinical response is defined as a 70-point decrease in CDAI score.
Time Frame: Baseline to Week 12
Population: All subjects who received at least one apheresis treatment session and had a CDAI score greater than 300 at baseline were included in the analysis population. The week 12 CDAI score was used for the analysis. Subjects without a week 12 CDAI score or subjects with a major violation on prohibited medications were considered a treatment failure.
Measure: Number; unit: percentage of participants
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 80 | 48
percentage of participants
  Baseline CDAI Score>300 | 43.8 | 27.1
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.0632, Fisher Exact
Statistical Analysis 2: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.0504, Fisher Exact (Mid-P-Value)

19. Post Hoc Outcome: Clinical Response in Subjects With a CDAI Score Less Than or Equal to 300
Description: A clinical response is defined as a 70-point decrease in CDAI score
Time Frame: Baseline to Week 12
Population: All subjects who received at least one apheresis treatment session and had a CDAI score less than or equal to 300 at baseline were included in the analysis population. The week 12 CDAI score was used for the analysis. Subjects without a week 12 CDAI score or with a major violation on prohibited medications were considered a treatment failure.
Measure: Number; unit: percentage of participants
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 77 | 30
percentage of participants | 39.0 | 43.3
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.8265, Fisher Exact

20. Post Hoc Outcome: Clinical Response Based on Previous Use of Tumor Necrosis Factor-Alpha (TNF-a) Inhibitors
Description: A clinical response is defined as a 70-point decrease in CDAI score
Time Frame: Baseline to Week 12
Population: All subjects who received at least one apheresis treatment session and previously used TNFa-inhibitors were included in the analysis population. The week 12 CDAI score was used for the analysis. Subjects without a week 12 CDAI score or subjects with a major violation on prohibited medications were considered a treatment failure.
Measure: Number; unit: percentage of participants
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 28 | 19
percentage of participants | 50.0 | 21.1
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.0676, Fisher Exact
Statistical Analysis 2: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.0506, Fisher Exact (Mid-P-Value)

21. Post Hoc Outcome: Clinical Response Based on No Previous Use of Tumor Necrosis Factor-Alpha (TNF-a) Inhibitors
Description: A clinical response is defined as a 70-point decrease in CDAI score
Time Frame: Baseline to Week 12
Population: All subjects who received at least one apheresis treatment session and who have not used TNFa-inhibitors were included in the analysis population. The week 12 CDAI score was used for the analysis. Subjects without a week 12 CDAI score or subjects with a major violation on prohibited medications were considered a treatment failure.
Measure: Number; unit: percentage of participants
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 129 | 59
percentage of participants | 39.5 | 37.3
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.8721, Fisher Exact

22. Post Hoc Outcome: Clinical Response Based on Use of 5-Aminosylisalates During the Study
Description: A clinical response is defined as a 70-point decrease in CDAI score
Time Frame: Baseline to Week 12
Population: All subjects who received at least one apheresis treatment session and who used 5-aminosylisalates during the study were included in the analysis population. The week 12 CDAI score was used for the analysis. Subjects without a week 12 CDAI score or subjects with a major violation on prohibited medication were considered a treatment failure.
Measure: Number; unit: percentage of participants
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 64 | 23
percentage of participants | 48.4 | 21.7
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.0289, Fisher Exact

23. Post Hoc Outcome: Clinical Response Based on no Use of 5-Aminosylisalates During the Study
Description: A clinical response is defined as a 70-point decrease in CDAI score
Time Frame: Baseline to Week 12
Population: All subjects who received at least one apheresis treatment session and who did not use 5-aminosylisalates during the study were included in the analysis population. The week 12 CDAI score was used for the analysis. Subjects without a week 12 CDAI score or subjects with a major violation on prohibited medications were considered a treatment failure.
Measure: Number; unit: percentage of participants
Arm/Group | Adacolumn | Sham
Number analyzed (Participants) | 93 | 55
percentage of participants | 36.6 | 38.2
Statistical Analysis 1: Comparison: Adacolumn vs Sham; Test type: Superiority or Other; p = 0.8618, Fisher Exact

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less